CLINICAL TRIAL: NCT01036126
Title: Automatic Versus Evaluative Components of Cue Reactivity
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903384; 03-DA-N384
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-08-19

CONDITIONS: Drug Dependence
Keywords: Nicotine; Cocaine; N-Back; Craving; Dependence
MeSH Terms: conditions — Substance-Related Disorders

SUMMARY:
Background:

- Relapse to drug abuse often happens in the presence of stimuli that are associated with previous drug use, also known as cues. Drug-taking behavior appears to be partly controlled by such cues. Some research suggests that cue-induced craving states are responsible for drug use and relapse, but other research suggests that cues can control drug taking without conscious craving or even awareness. Researchers are interested in using functional magnetic resonance imaging (fMRI) to study how individuals respond to drug-related cues and how these cues affect craving on a conscious or unconscious level.

Objectives:

- To determine how drug-related stimuli (cues) affect thinking, information processing, and body reactions in current drug users.

Eligibility:

- Individuals between 18 and 50 years of age who are dependent on either tobacco or crack-cocaine, or are healthy volunteers who are not dependent on either drug.

Design:

* The study will require two sessions, a training session and a testing session, that will take place within 48 hours of each other. Between the two test sessions, participants may not consume alcohol, tobacco, or illegal drugs, and must restrict caffeine consumption.
* During the first session, participants will complete questionnaires about tobacco/cocaine use and craving, and will be trained on the tasks to be performed in the MRI scanner.
* During the second session, participants will perform concentration tasks and look at pictures, some of which will be tobacco/cocaine related. Body reactions such as heart rate, pupil dilation, and sweating will be measured during this session. Some participants will have actual MRI scanning, while others will have mock MRI scanning.
* After the MRI session, participants will complete questionnaires about craving and responses to the scan.

DETAILED DESCRIPTION:
Relapse to drug abuse often happens in the presence of stimuli that are associated with previous drug-use, and drug-taking behavior appears to be partly controlled by such cues. While some theories postulate that such facilitation is mediated by cue-induced craving states, others hypothesize that the underlying processes are highly automatized and can happen without conscious control or even awareness. One way to approach psychological mechanisms of cue reactivity is to measure disruption of ongoing mental activity by drug-related material in dependent individuals while manipulating the degree to which cognitive evaluative processes can unfold. Craving measurement under these conditions can elucidate its relationship with automatic processing versus conscious evaluation of drug cues. Autonomic and neural correlates can be identified by concomitant psychophysiological and fMRI recording. Results from these studies will shed light on the role of spontaneous automatic reactions versus cognitive evaluation for different measures of cue reactivity. By helping to elucidate the psychological mechanisms and neurobiological basis of drug-cue reactivity in dependent individuals, this may have substantial implications for the understanding of mechanisms and treatment of drug dependence. Thus, while there are no direct benefits to subjects participating in these experiments, the results may benefit the health of society. MRI-related risks to subjects (injury from metal implants, claustrophobia, temporary deafness due to the loud banging noises) will be minimized by prescreening and providing earplugs. Drug-related cues may induce acute craving; subjects will be dismissed only after craving levels have returned to baseline.

ELIGIBILITY:
* INCLUSION CRITERIA:

Smokers:

Regular smoking of greater than or equal to 20 cigarettes other than ultra-low nicotine cigarettes per day for at least two years. Experienced withdrawal signs after not smoking for several hours. Score on the Fagerstrom Test for Nicotine Dependence greater than or equal to 3.

No intention to quit or reduce tobacco use, and no treatment for tobacco dependence currently or during the previous 3 months.

No history of abuse of or dependence to any other drug.

Age at least 18 and not older than 50 years.

Controls:

Smoked less than 5 cigarettes during lifetime

No history of abuse of or dependence to any drug, including alcohol.

Age at least 18 and not older than 50 years.

Cocaine abusers:

Reported regular crack-cocaine use for at least six months. Meeting DSM-IV criteria for cocaine dependence.

No intention to quit or reduce cocaine use, and no treatment for cocaine dependence currently or during the previous 3 months.

No dependence on any other drug except nicotine. Recreational use of other drugs of abuse without meeting dependence criteria is not an exclusion criterion.

Age at least 18 and not older than 50 years.

Controls:

No history of dependence on any drug except nicotine.

Age at least 18 and not older than 50 years.

EXCLUSION CRITERIA: All subject groups

Female subjects: pregnancy (a urine pregnancy test will be performed before each MRI experimental session).

Presence of metal objects in the body (e.g. some artificial joints, bone pins, surgical clips, skull plate, dental braces) or implanted electronic devices (e.g. cardiac pacemaker, neurostimulator)

Claustrophobia.

For experiments involving MRI, left-handed or ambidextrous as determined by the Edinburgh Handedness Inventory.

Cardiovascular or cerebrovascular diseases.

Major psychiatric disorders including mood, anxiety or psychotic disorders.

History of or current neurological illnesses including seizure disorders, migraine, multiple sclerosis, movement disorders, head trauma, CVA or CNS tumor. Gross structural brain abnormalities as revealed by T1 weighted images. Use of medication that may affect the CNS at the time of scanning (e.g. b-blocker or analgesics).

Learning disability, amnesia or other conditions that impede memory and attention. IQ less than 85.

HIV-positivity.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2003-08-12; Study Completion 2010-08-19

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

REFERENCES:
- [Background] Abrams DB, Monti PM, Carey KB, Pinto RP, Jacobus SI. Reactivity to smoking cues and relapse: two studies of discriminant validity. Behav Res Ther. 1988;26(3):225-33. doi: 10.1016/0005-7967(88)90003-4. No abstract available. PMID 3408457
- [Background] Bagby RM, Parker JD, Taylor GJ. The twenty-item Toronto Alexithymia Scale--I. Item selection and cross-validation of the factor structure. J Psychosom Res. 1994 Jan;38(1):23-32. doi: 10.1016/0022-3999(94)90005-1. PMID 8126686
- [Background] Baker TB, Morse E, Sherman JE. The motivation to use drugs: a psychobiological analysis of urges. Nebr Symp Motiv. 1986;34:257-323. PMID 3627296